CLINICAL TRIAL: NCT07399665
Title: Open-label Single-arm, Non-interventional, Multi-centre Study for Evaluation of Clinical and Patient Reported Outcomes in Adult Patients With CRSwNP on Tezepelumab
Brief Title: ReAl-woRld Evaluation of tEzepelumab for Chronic rhinoSinusitis With Nasal Polyps in Russia
Acronym: ARES
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5242R00010
Record Dates: First submitted 2025-11-24; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps (CRSwNP); Asthma
Keywords: Tezepelumab; CRSwNP
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ARES is a multi-centre, retrospective-prospective, non-comparative and non-interventional (observational) cohort study involving primary and secondary data collection within real-world settings of participants who have initiated tezepelumab (no more than 4 weeks before inclusion) for treatment of CRSwNP (with or without comorbid asthma).

DETAILED DESCRIPTION:
ARES is a multi-centre, retrospective-prospective, non-comparative and non-interventional (observational) cohort study involving primary and secondary data collection within real-world settings of participants who have initiated tezepelumab (no more than 4 weeks before inclusion) for treatment of CRSwNP (with or without comorbid asthma) to capture real-world data on the effectiveness and use patterns of tezepelumab outside the controlled conditions of a randomized clinical trial.

The study will be conducted in real-world setting at approximately 10 sites in the Russian Federation. A total of 110 eligible adult participants (aged ≥18 years) of both sexes who will be treated with tezepelumab as prescribed by their treating physicians will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 18 years or older at the time of signing the ICF.
2. Diagnosis of CRSwNP established for at least 52 weeks prior to tezepelumab initiation.
3. Availability of participants' medical records for at least 52 weeks prior to tezepelumab initiation, including history of sCS use / nasal polyps surgery (or information about contraindications / intolerance to).
4. Prescribed and initiated treatment with tezepelumab according to SmPC and local market reimbursement criteria. A period between treatment initiation and enrolment should be no more than 4 weeks.
5. The severity of CRSwNP consistent with need for surgery as defined by total NPS ≥ 5 (at least 2 for each nostril) at the enrollment.
6. Nasal Blockage score as part of SNOT-22 (NBS-SNOT-22) ≥ 3 at the enrollment.
7. SNOT-22 total score ≥ 30 at enrollment or up to 12 weeks before enrollment.
8. Currently receive care from specialist physicians (e.g., otolaryngologist) at the Investigator's or sub-Investigator's site.
9. Provision of signed and dated written informed consent.
10. Participants are able to read, understand and complete the questionnaires required by the protocol.

Exclusion Criteria:

1. Any contraindication to tezepelumab as per the approved product SmPC in Russia or in the opinion of the Investigator.
2. Administration of concurrent biologic drug for CRSwNP / asthma since the index date, except for stable allergen immunotherapy (defined as a stable dose and regimen at the time of enrolment). Enrolment of patients who were switched from other biologic(s) to tezepelumab is allowed, and an acceptable timeframe since the last prior biologic drug is ≥ 60 days. The number of participants with prior biologic treatment (switching to tezepelumab) should be targeted at 20% or less.
3. Participation in an observational study that might, in the Investigator's opinion, influence the assessment for the current study, or participation in an interventional clinical trial in the last 3 months.
4. Pregnancy or lactation period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants of both sexes aged 18 years and older with severe nasal polyposis (NPS ≥ 5) and the need for surgery, severe nasal congestion (Nasal Blockage ≥ 3 as part of SNOT-22), significant decrease in quality of life (SNOT-22 ≥ 30) despite the use of intranasal CS, who have indications for the prescription of biological therapy, who have commenced treatment with Tezepelumab as determined by their routine clinical care, will be enrolled in the otolaryngology setting of clinical institutions in Russia. Eligible patients will be enrolled consecutively at each site to minimize selection bias at each site. The study will target to enroll no more than 20% participants switching from a prior biologic drug to Tezepelumab and no more than 60% participants with comorbid asthma.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-12-25 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
1. Change in endoscopic status of CRSwNP based on NPS | time points to measure: baseline and at Weeks 4, 24 and 52 following tezepelumab initiation
  Change in NPS score from baseline
2. Change in a nasal congestion status based on Nasal Blockage score as part of SNOT-22 (NBS-SNOT-22) | time points to measure: baseline and at Weeks 4, 24 and 52 following tezepelumab initiation
  Change in Nasal blockage score as part of SNOT-22 (NBS-SNOT-22) from baseline
3. Change in endoscopic status of CRSwNP based on NPS | time points to measure: baseline and at Weeks 4, 24 and 52 following tezepelumab initiation
  Proportion of patients with at least a 1-point improvement in NPS score from baseline
4. Change in a nasal congestion status based on Nasal Blockage score as part of SNOT-22 (NBS-SNOT-22) | time points to measure: baseline and at Weeks 4, 24 and 52 following tezepelumab initiation
  Proportion of patients with at least a 1-point improvement in Nasal blockage score as part of SNOT-22 (NBS-SNOT-22) from baseline

SECONDARY OUTCOMES:
1. Change in SNOT-22 total score from baseline | time points to measure: baseline and at Weeks 4, 24 and 52 following tezepelumab initiation
  To describe the participant-reported evaluation of the symptoms of CRSwNP using the Sinonasal Outcome Test-22 (SNOT-22) at baseline* and up to 52 weeks following tezepelumab initiation.
2. Proportion of participants with clinically meaningful change (reduction in SNOT-22 score by ≥ 8.9) from baseline | To describe the participant-reported evaluation of the symptoms of CRSwNP using the Sinonasal Outcome Test-22 (SNOT-22) at baseline* and up to 52 weeks following tezepelumab initiation.
  To describe the participant-reported evaluation of the symptoms of CRSwNP using the Sinonasal Outcome Test-22 (SNOT-22) at baseline* and up to 52 weeks following tezepelumab initiation.
3. Change in loss of smell (as a part of SNOT-22) from baseline | time points to measure: baseline and at Weeks 4, 24 and 52 following tezepelumab initiation
  To describe a smell status based on loss of smell score as part of SNOT-22 at baseline* and up to 52 weeks following tezepelumab initiation.
4. Proportion of patients with at least a 1-point change in loss of smell (as a part of SNOT-22) from baseline | time points to measure: baseline and at Weeks 4, 24 and 52 following tezepelumab initiation
  To describe a smell status based on loss of smell score as part of SNOT-22 at baseline* and up to 52 weeks following tezepelumab initiation.
5. Change in Lund-Mackay score from baseline | time points to measure: baseline and at Weeks 4, 24 and 52 following tezepelumab initiation
  To describe status of nasal cavity and paranasal sinuses using CT and Lund-Mackay score at baseline* and up to 52 weeks following tezepelumab initiation.
6. Change in ACQ-5 score from baseline | time points to measure: baseline and at Weeks 4, 24 and 52 following tezepelumab initiation
  To describe asthma control questionnaire (ACQ-5) among participants with ongoing diagnosis of asthma
7. Proportion of participants with ACQ-5 response (reduction of ≥ 0.5 in score from baseline) | time points to measure: baseline and at Weeks 4, 24 and 52 following tezepelumab initiation
  To describe asthma control questionnaire (ACQ-5) among participants with ongoing diagnosis of asthma
8. Number (proportion) of participants with CRSwNP-related healthcare resource utilisation (by each type) | time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  To describe CRSwNP-related healthcare resource utilisation (HCRU)
9. Annualised rates of CRSwNP-related hospitalisation, emergency calls (or emergency department visits), and unscheduled out-patient visits to a physician | time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  To describe CRSwNP-related healthcare resource utilisation (HCRU)
10. Annualised rates of CRSwNP-related scheduled physician visits or healthcare calls for CRSwNP | time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  To describe CRSwNP-related healthcare resource utilisation (HCRU).
11. Median overall duration (days) of CRSwNP-related hospitalisations | time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  To describe CRSwNP-related healthcare resource utilisation (HCRU)
12. Number (proportion) of participants with asthma-related healthcare resource utilisation (by each type) | time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  To describe asthma-related HCRU among participants with ongoing diagnosis of asthma
13. Annualised rates of asthma-related hospitalisation, emergency calls (or emergency department visits), and unscheduled out-patient visits to a physician | time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  To describe asthma-related HCRU among participants with ongoing diagnosis of asthma
14. Annualised rates of asthma-related scheduled physician visits or healthcare calls for asthma | time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  To describe asthma-related HCRU among participants with ongoing diagnosis of asthma
15. • Median overall duration (days) of asthma-related hospitalisations | time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  To describe asthma-related HCRU among participants with ongoing diagnosis of asthma
16. Annualised rate of CRSwNP exacerbations | time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  To describe CRSwNP exacerbations.
17. Change in annualised rate of CRSwNP exacerbations from the baseline period to the follow-up period after tezepelumab initiation | time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  To describe CRSwNP exacerbations.
18. Proportion of participants with 0, 1, 2, ≥3 CRSwNP exacerbations | time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  To describe CRSwNP exacerbations.
19. Cumulative days of CRSwNP exacerbations (calculated in participants who had CRSwNP exacerbations at baseline) | time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  To describe CRSwNP exacerbations.
20. Annualised rate of severe* asthma exacerbations | time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  To describe severe asthma exacerbations among participants with ongoing diagnosis of asthma.
21. Change in annualised rate of severe* asthma exacerbations from the baseline period to the follow-up period after tezepelumab initiation | time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  To describe severe asthma exacerbations among participants with ongoing diagnosis of asthma.
22. Proportion of participants with 0, 1, 2, ≥3 severe* asthma exacerbations | time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  To describe severe asthma exacerbations among participants with ongoing diagnosis of asthma.
23. Cumulative days of severe* asthma exacerbations (calculated in participants who had asthma exacerbations at baseline) | time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  To describe severe asthma exacerbations among participants with ongoing diagnosis of asthma.
24. Median duration (days) of treatment with tezepelumab (to be calculated in all enrolled participants) | time points to measure: Week 52/End of Study
  To describe tezepelumab treatment features, including duration of therapy, in the 52 weeks following initiation of treatment.
25. Proportion of participants with tezepelumab discontinuation overall and by reason | time points to measure: Week 52/End of Study
  To describe tezepelumab treatment features, including duration of therapy, discontinuation, and reasons for discontinuation in the 52 weeks following initiation of treatment.
26. • Median time (days) to tezepelumab discontinuation (to be calculated in participants who discontinued tezepelumab earlier than Week 52 by any reason) | time points to measure: Week 52/End of Study
  To describe tezepelumab treatment features, including duration of therapy, discontinuation, and reasons for discontinuation in the 52 weeks following initiation of treatment.
27. Proportion of participants discontinued tezepelumab and switched to other biologic drug for CRSwNP / asthma treatment and reason(s) | time points to measure: Week 52/End of Study
  To describe duration of Tezepelumab therapy in the 52 weeks following initiation of treatment.
28. Change in blood eosinophils level (cells/μL) from baseline | time points to measure: baseline and at Weeks 4, 24 and 52 following tezepelumab initiation
  To describe biomarkers profile of participants and its dynamics from baseline* and up to 52 weeks following tezepelumab initiation.
29. Change in total IgE level (IU/mL) from baseline | time points to measure: baseline and at Weeks 4, 24 and 52 following tezepelumab initiation
  To describe biomarkers profile of participants and its dynamics from baseline* and up to 52 weeks following tezepelumab initiation.
30. Mean duration (days) of treatment with tezepelumab (to be calculated in all enrolled participants) | time points to measure: Week 52/End of Study
  To describe tezepelumab treatment features, including duration of therapy in the 52 weeks following initiation of treatment.
31. Proportion of participants discontinued tezepelumab and switched to other biologic drug for CRSwNP / asthma treatment and reason(s) | time points to measure: Week 52/End of Study
  To describe reasons for discontinuation in the 52 weeks following initiation of treatment.

OTHER OUTCOMES:
1. Proportion of participants with medications for CRSwNP treatment by drug class | time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  To describe use of CRSwNP treatment (including surgery) at baseline* and up to 52 weeks following tezepelumab initiation.
2. Proportion of patients with InCS use | time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  To describe use of CRSwNP treatment (including surgery) at baseline* and up to 52 weeks following tezepelumab initiation.
3. Mean daily dose of sCS (to be calculated in participants who used sCS) | time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  To describe use of CRSwNP treatment (including surgery) at baseline* and up to 52 weeks following tezepelumab initiation.
4. Proportion of patients with oral antibiotics use due to CRSwNP or its exacerbation | time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  To describe use of CRSwNP treatment (including surgery) at baseline* and up to 52 weeks following tezepelumab initiation.
5. Proportion of patients with any sCS use due to CRSwNP or its exacerbation ('systemic' means oral, parenteral CS) | time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  To describe use of CRSwNP treatment (including surgery) at baseline* and up to 52 weeks following tezepelumab initiation.
6. Proportion of patients with 0, 1 and ≥2 courses of sCS due to CRSwNP or its exacerbation | time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  To describe use of CRSwNP treatment (including surgery) at baseline* and up to 52 weeks following tezepelumab initiation.
7. Median number of sCS courses due to CRSwNP or its exacerbation | time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  To describe use of CRSwNP treatment (including surgery) at baseline* and up to 52 weeks following tezepelumab initiation.
8. • Proportion of patients with any other biologic therapy use due to CRSwNP and/or severe asthma | time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  To describe use of CRSwNP treatment (including surgery) at baseline* and up to 52 weeks following tezepelumab initiation.
9. Medication possession ratio (MPR) - total days' supply of a medication in a particular time period, divided by the number of days in the time period | time points to measure: Week 52/End of Study
  To describe use of CRSwNP treatment (including surgery) at baseline* and up to 52 weeks following tezepelumab initiation.
10. Proportion of participants with CRSwNP-related surgical interventions by type of surgery | time points to measure: from the date of CRSwNP diagnosis and up to 52 weeks following tezepelumab initiation
  To describe use of CRSwNP treatment (including surgery) at baseline* and up to 52 weeks following tezepelumab initiation.
11. Median time since the most recent nasal polyp surgery, calculated at the date of tezepelumab initiation. | The date of tezepelumab initiation
  To describe use of CRSwNP treatment (including surgery) at baseline* and up to 52 weeks following tezepelumab initiation.
12. Proportion of patients with 0, 1, 2, 3, 4 and ≥5 CRSwNP-related surgical interventions | time points to measure: from the date of CRSwNP diagnosis and up to 52 weeks following tezepelumab initiation
  To describe use of CRSwNP treatment (including surgery) at baseline* and up to 52 weeks following tezepelumab initiation.
13. Median number of CRSwNP-related surgical interventions | time points to measure: from the date of CRSwNP diagnosis and up to 52 weeks following tezepelumab initiation
  To describe use of CRSwNP treatment (including surgery) at baseline* and up to 52 weeks following tezepelumab initiation.
14. Proportion of patients with indications for CRSwNP-related surgery | time points to measure: from the index date and up to 52 weeks following tezepelumab initiation
  To describe the need for sCS use and/or nasal polyp surgery during the tezepelumab treatment period (52 weeks).
15. Proportion of patients with the need of sCS therapy | time points to measure: from the index date and up to 52 weeks following tezepelumab initiation
  To describe the need for sCS use and/or nasal polyp surgery during the tezepelumab treatment period (52 weeks).
16. Median time to first sCS use and/or nasal polyp surgery during the treatment period | time points to measure: from the index date and up to 52 weeks following tezepelumab initiation
  To describe the need for sCS use and/or nasal polyp surgery during the tezepelumab treatment period (52 weeks).
17. Patients' adherence to treatment, which will be calculated at the date of the corresponding visit as (actual number of injections received / planned number of injections prescribed by physician * 100%) | time points to measure: baseline and at Weeks 4, 24 and 52 following tezepelumab initiation
  To describe participants' adherence to treatment up to 52 weeks following tezepelumab initiation.
18. Proportion of participants with each category of PGI-S scale | time points to measure: baseline
  To describe patient-reported impression of disease severity (PGI-S) scale
19. • Proportion of participants with each category of PGI-C scale | time points to measure: Weeks 4, 24 and 52 following tezepelumab initiation
  To describe patient-reported impression of treatment using Patient Global Impression of Change (PGI-C) scale throughout the 52-week treatment period.
20. Proportion of participants with CRSwNP-related surgical interventions by volume of surgery | time points to measure: from the date of CRSwNP diagnosis and up to 52 weeks following tezepelumab initiation
  To describe use of CRSwNP treatment (including surgery) at baseline* and up to 52 weeks following tezepelumab initiation.

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - ARES, Moscow
  - ARES, Ryazan
  - ARES, Saint-Petesburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/